CLINICAL TRIAL: NCT00623506
Title: Adjunctive Pregnenolone in Veterans With Mild TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Durham VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VA IRB# 01209; VA IRB# 01209
Record Dates: First submitted 2008-02-15; First posted 2008-02-26 (Estimated); Results first posted 2013-06-20 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-05

CONDITIONS: Traumatic Brain Injury
Keywords: TBI; Pregnenolone; Cognition
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Pregnenolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): Pregnenolone
  Interventions: Drug: Pregnenolone
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregnenolone — Placebo for two weeks (during placebo lead-in), then:
  Pregnenolone 100 mg in divided doses (50 mg, PO, BID) Pregnenolone 300 mg in divided doses (150 mg, PO, BID) Pregnenolone 500 mg in divided doses (250 mg, PO, BID)
  Arms: 1
Drug: Placebo — Placebo for two weeks (placebo lead in), then:
  Placebo equivalent to Pregnenolone arm: 100 mg in divided doses (50 mg, PO, BID) Placebo equivalent to Pregnenolone arm: 300 mg in divided doses (150 mg, PO, BID) Placebo equivalent to Pregnenolone arm: 500 mg in divided doses (250 mg, PO, BID)
  Arms: 2

SUMMARY:
Mild traumatic brain injury (TBI) is common among veterans who have served in OEF/OIF (Operation Enduring Freedom in Afghanistan/Operation Iraqi Freedom) and other theatres. Delayed symptoms may occur following TBI, including cognitive symptoms (impaired attention, processing speed, executive functioning), as well as behavioral symptoms such as anxiety, depression, and irritability (Fann et al. 2004; Holsinger et al. 2002). Neuroactive steroids have neuroprotective effects in rodent models of TBI (Djebaili et al. 2005; Djebaili et al. 2004; He et al. 2004; Pettus et al. 2005; Roof et al. 1997) and the neuroactive steroid pregnenolone and its sulfated derivative also markedly enhance learning and memory in rats (Akwa et al. 2001; Flood et al. 1992; Flood et al. 1995; Vallee et al. 1997; Vallee et al. 2003). In humans, reductions in pregnenolone (George et al. 1994) and its GABAergic metabolite allopregnanolone (Uzunova et al. 1998) have been associated with depressive symptoms. Pharmacological intervention with the neuroactive steroid pregnenolone could therefore result in a multi-targeted treatment approach, potentially improving cognitive deficits as well as anxiety and depression symptoms following TBI.

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
Inclusion Criteria:

1. 18-55 years of age, any ethnic group, either sex
2. History of mild TBI since September 2001. TBI occurring at age 18 or older.
3. We will adhere to the operational definition of mild TBI suggested by the World Health Organization Task Force (Holm et al.2005), with the exception of the Glasgow Coma Scale Score criteria (not available for these participants).
4. Ability to participate fully in the informed consent process.
5. No anticipated need to alter medications for the 10-week duration of the study.

Exclusion Criteria:

1. For this pilot study, we will exclude patients who report a history of seizures.
2. Serious unstable medical illness. History of cerebrovascular accident, prostate, uterine, or breast cancer. Use of oral contraceptives or other hormonal supplementation such as estrogen.
3. Current active suicidal and/or homicidal ideation, intent or plan.
4. Concomitant medications for medical conditions will be addressed on a case-by-case base and determined if exclusionary.
5. Current DSM-IV (Diagnostic and Statistical Manual, Fourth Edition) diagnosis of bipolar disorder, schizophrenia or other psychotic disorder, or cognitive disorder due to a general medical condition other than TBI.
6. Female patients who are pregnant or breast-feeding.
7. Known allergy to study medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2008-01; Primary Completion 2009-08 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine E Marx, MD, MA, Principal Investigator — Durham VAMC
Locations (1):
- Durham VA Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the Durham Medical Center, Durham, NC.
Pre-assignment Details: Each subject received a two week placebo-lead in following enrollment.
Groups:
- Pregnenolone: Pregnenolone
  Pregnenolone : Pregnenolone 100 mg in divided doses (50 mg, PO, BID) Pregnenolone 300 mg in divided doses (150 mg, PO, BID) Pregnenolone 500 mg in divided doses (250 mg, PO, BID)
- Placebo: Placebo
  Subjects received placebo study medication; dispensed exactly as active study medication was dispensed.
Period: Overall Study
Arm/Group | Pregnenolone | Placebo
Started | 15 | 15
Week 4 | 11 | 11
Completed | 11 | 11
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregnenolone | Placebo | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 34.27 (10.51) | 36.38 (9.74) | 35.76 (9.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 9 | 10 | 19
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Brief Assessment of Cognition in Affective Disorders (BAC-A)
Description: Mean change scores (Week 2 minus Week 10) to assess cognitive changes. The BAC-A includes brief assessments of executive functions, verbal fluency, attention, verbal memory, working memory and motor speed. Z-scores are calculated from composite scores. Higher z-scores are indicative of better cognitive performance, lower z-scores are indicative of lower cognitive performance. Range of z-scores anticipated to be between -3 and 3. Mean change scores from week 2 and week 10 (Week 2 minus Week 10).
Time Frame: Week 2, Week 10
Population: 22 out of 30 patients randomized completed 4 or more weeks of the study and were retained for data analysis. Statistics were completed using Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 11 | 11
units on a scale | 0.61 (0.14) | 0.80 (0.17)

2. Secondary Outcome: Clinician Administered PTSD Scale (CAPS)
Description: Mean change scores (Week 2 minus Week 10) in posttraumatic stress disorder symptoms. Scores may range from 0 (no symptoms) to 136 (severe symptoms; score of 136 is based on the first 17 CAPS items administered).
  A reduced CAPS score indicates a reduction in (improvement) PTSD symptoms, while an increase in CAPS score indicates an increase (worsening) in PTSD symptoms.
Time Frame: Week 2, Week 10
Population: 22 out of 30 patients randomized completed 4 or more weeks of the study and were retained for data analysis. Statistics were completed using LOCF.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 11 | 11
units on a scale | -8.5 (3.22) | -7.3 (4.74)

3. Secondary Outcome: Quick Inventory of Depressive Symptomatology (QIDS)
Description: The QIDS total scores range from 0 to 27. Total score is obtained by adding the scores for each of the nine symptom domains of the DSM-IV Major Depressive Disorder (MDD) criteria: depressed mood,loss of interest or pleasure,concentration/decision making,self-outlook,suicidal ideation, energy/fatigability,sleep,weight/appetite change,and psychomotor changes. Each item is rated 0-3 (0=least or no severity, 3=greatest severity).
Time Frame: Week 2, Week 10
Population: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Pregnenolone | Placebo
Number analyzed (Participants) | 11 | 11
units on a scale | -1.09 (0.73) | -0.54 (0.71)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected following the one-week placebo-lead phase and at each subsequent study visit and telephone check-in. Adverse events were collected during 11 out of the 12 weeks.
Arm/Group | Pregnenolone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 6/11 | 6/11
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pregnenolone (N=11) | Placebo (N=11)
Headache (General disorders) | 3 (4) | 1 (1) — Hillside Adverse Event Scale
Excitation and Agitation (General disorders) | 1 (1) | 0 (0) — Hillside Adverse Event Scale
Restlessness (General disorders) | 0 (0) | 1 (1) — Hillside Adverse Event Scale
Increased motor activity (General disorders) | 0 (0) | 1 (1) — Hillside Adverse Event Scale
Decreased Motor Activity (General disorders) | 0 (0) | 1 (2) — Hillside Adverse Event Scale
Malaise (General disorders) | 1 (1) | 1 (1) — Hillside Adverse Event Scale
Insomnia (General disorders) | 0 (0) | 1 (2) — Hillside Adverse Event Scale
Hypersomnia (General disorders) | 1 (1) | 0 (0) — Hillside Adverse Event Scale
Drowsiness (General disorders) | 1 (1) | 3 (7) — Hillside Adverse Event Scale
Cramps (General disorders) | 0 (0) | 1 (1) — Hillside Adverse Event Scale
Akathisia (General disorders) | 0 (0) | 1 (1) — Hillside Adverse Event Scale
Dizziness (General disorders) | 1 (1) | 1 (1) — Hillside Adverse Event Scale
Dry Mouth (General disorders) | 1 (1) | 1 (1) — Hillside Adverse Event Scale
Blurred Vision (General disorders) | 0 (0) | 1 (1) — Hillside Adverse Event Scale
Constipation (General disorders) | 0 (0) | 1 (1) — Hillside Adverse Event Scale
Nausea (General disorders) | 1 (1) | 1 (1) — Hillside Adverse Event Scale
Decreased Interest in Sex (General disorders) | 1 (2) | 0 (0) — Hillside Adverse Event Scale
Impaired Sexual Performance (General disorders) | 1 (1) | 1 (1) — Hillside Adverse Event Scale
Dermatological (General disorders) | 2 (4) | 2 (4) — Hillside Adverse Event Scale
Muscle pain/stiffness (General disorders) | 1 (1) | 0 (0) — Hillside Adverse Event Scale
Decreased Appetite (General disorders) | 1 (1) | 0 (0) — Hillside Adverse Event Scale
Increased appetite (General disorders) | 1 (1) | 2 (4) — Hillside Adverse Event Scale

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes